CLINICAL TRIAL: NCT05690932
Title: A Single-Dose, Open-Label, Two-Part, Randomized, Crossover Formulation Bridging and Food Effect Study to Assess the Effect of Formulation and Food on the Absorption and Bioavailability of PBI-200 in Normal Healthy Volunteers
Brief Title: A Formulation Bridging and Food Effect Study of PBI-200 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pyramid Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PBI-200-105
Record Dates: First submitted 2023-01-10; First posted 2023-01-19 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Formulation Bridging; Food Effect

STUDY DESIGN:
Intervention Model Description: Single-dose, open-label, randomized, three-way crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Capsule (Experimental): Study drug will be administered with water after an overnight fast.
  Interventions: Drug: PBI-200 Capsule
- Tablet (Experimental): Study drug will be administered with water after an overnight fast.
  Interventions: Drug: PBI-200 Tablet
- Suspension (Experimental): Study drug will be administered with water after an overnight fast.
  Interventions: Drug: PBI-200 Suspension
- Fasted (Experimental): Study drug will be administered with water after an overnight fast.
  Interventions: Drug: PBI-200 Tablet
- Low-fat Meal (Experimental): Study drug will be administered with water after an overnight fast, after which time a standard low-fat breakfast will be given.
  Interventions: Drug: PBI-200 Tablet
- High-fat Meal (Experimental): Study drug will be administered with water after an overnight fast, after which time a standard high-fat breakfast will be given.
  Interventions: Drug: PBI-200 Tablet

INTERVENTIONS:
Drug: PBI-200 Tablet — Single dose of PBI-200 tablet
  Arms: Fasted; High-fat Meal; Low-fat Meal; Tablet
Drug: PBI-200 Capsule — Single dose of PBI-200 capsule
  Arms: Capsule
Drug: PBI-200 Suspension — Single dose of PBI-200 suspension
  Arms: Suspension

SUMMARY:
This is a single-dose, two-part, crossover formulation bridging and food effect study to assess the effect of formulation and food on the absorption and bioavailability of PBI-200 in normal, healthy volunteers.

DETAILED DESCRIPTION:
This is a single-dose, two-part crossover formulation bridging (Part A) and tablet food effect (Part B) study in normal, healthy volunteers. Part A will be conducted to evaluate the pharmacokinetics (PK) and relative bioavailability of 3 formulations of PBI-200; each volunteer will serve as their own control. In Part B, PBI-200 tablets will be dosed under fasting and fed (low-fat and high-fat meals) conditions to evaluate the effect of food on the PK of PBI-200.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant, non-lactating female between 18 and 55 years of age (inclusive).
* Body Mass Index (BMI) between 18.0 and 32.0 kg/m² (inclusive).
* Non-smoking/non-vaping, healthy, with no history of clinically relevant medical illness.

Exclusion Criteria:

* History or presence of clinically significant cardiovascular, pulmonary, respiratory, hepatic, renal, hematological, gastrointestinal, endocrine, immunologic, dermatologic, neurological, or psychiatric disease which, in the opinion of the Investigator, would jeopardize the safety of the volunteer or impact the validity of the study results.
* History of gastrointestinal/hepatobiliary or other surgery that may affect PK profiles (i.e., hepatectomy, gastric, bypass, or digestive organ resection).
* Intolerance to repeated venipuncture.
* Smoking or use of tobacco products (including vaping) within 3 months prior to the first study drug administration.
* Have a positive drug/alcohol screen, or history or presence of alcoholism or drug abuse within 6 months of first study drug administration.
* Volunteers with a corrected QT using Fridericia's formula (QTcF) prolongation over 450 milliseconds at Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2022-02-24 (Actual); Primary Completion 2022-05-23 (Actual); Study Completion 2022-05-23 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration [C(max)] of PBI-200 | 8 days
  Maximum (peak) plasma drug concentration
Area Under the Concentration-Time Curve (AUC) of PBI-200 from time zero to the time of th last measurable concentration [AUC(0-t)] | 8 days
  AUC, calculated using linear up / log down trapezoidal method from time zero to time t, where t is the time of the last measurable concentration.
AUC of PBI-200 from time zero to infinity [AUC(0-inf)] | 8 days
  AUC from time zero to infinity, AUC(0-inf) = AUC(0-t) + Ct/kel, where kel is the terminal rate constant and Ct is the last measurable concentration.

SECONDARY OUTCOMES:
Time to Maximum Concentration [T(max)] of PBI-200 | 8 days
  T(max) will be determined from the observed plasma concentration data
Terminal elimination half-life [T(1/2)] | 8 days
  Apparent terminal elimination half-life, calculated as ln(2)/kel
Incidence, frequency and severity of adverse events (AEs) | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Pyramid Biosciences
Locations (1):
- Bio-Kinetic Clinical Applications, Springfield, Missouri, United States

IPD SHARING:
Plan to Share IPD: No